CLINICAL TRIAL: NCT04999800
Title: A Prospective Clinical Study to Evaluate the Efficacy and Safety of Pembrolizumab Combined With Anlotinib in First-line Treatment for Patients With of R/M HNSCC PD-L1 CPS≥1
Brief Title: Study of Pembrolizumab Combined With Anlotinib in the First Line Therapy for R/M HNSCC With CPS≥1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shi Yuankai (Unknown)
Responsible Party: Sponsor-Investigator, Shi Yuankai, Director, Head of Oncology, Chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCT20217
Record Dates: First submitted 2021-07-12; First posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and Neck Cancer; immune therapy; Pembrolizumab combined with Anlotinib
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — pembrolizumab; anlotinib

STUDY DESIGN:
Intervention Model Description: Pembrolizumab combined with Anlotinib
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab combined with Anlotinib (Experimental): Anlotinib 12 mg QD p.o for 2 weeks and then stop for 1 week, combined with Pembrolizumab 200 mg iv on day 1, and every 21 days is a treatment cycle until the disease progresses or the toxicity cannot be tolerated
  Interventions: Drug: Pembrolizumab; Drug: Anlotinib

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab (formerly lambrolizumab, brand name Keytruda) is a humanized antibody used in cancer immunotherapy. This includes to treat melanoma, lung cancer, head and neck cancer, Hodgkin lymphoma, an stomach cancer
  Other Names: Keytruda
Drug: Anlotinib — Anlotinib is an oral small molecule multi-target receptor tyrosine kinase inhibitor
  Other Names: AL3818

SUMMARY:
This trial is main evaluate the efficacy and safety of Pembrolizumab combined with Anlotinib in the first-line treatment of recurrent or metastatic head and neck squamous cell carcinoma with CPS≥1

DETAILED DESCRIPTION:
This test is a single-center, prospective phase II clinical research, plan included in 20 cases of eligible subjects, assessment in China PD-L1 CPS≥1 or more recurrent and/or metastatic head and neck squamous cell carcinoma patients, Pembrolizumab combined with Anlotinib for the initial curative effect, adverse reaction and safety, provide the basis for subsequent clinical trials

ELIGIBILITY:
Inclusion Criteria:

* 1) Voluntarily sign written informed consent before screening; 2) Age ≥18 years old; 3) ECOG physical status score 0-1; 4) Histologically or cytologically confirmed squamous cell carcinoma of the head and neck (HNSCC) with primary site of oral cavity, oropharynx, hypopharynx or larynx; 5) Recurrent and/or metastatic HNSCC without indications of local radical treatment; 6) According to the efficacy evaluation criteria for solid tumors (RECIST version 1.1), at least one measurable lesion can be selected as the target lesion after receiving previous radiotherapy only if there has been definite disease progression 3 months after the end of radiotherapy; 7) Sufficient tumor tissue samples for PD-L1 immunohistochemical detection; 8) Expected survival of more than 3 months; 9) The main organs function normally, that is, they meet the following criteria: I. Blood routine (no blood transfusion, erythropoietin (EPO), granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) treatment within 14 days before screening examination) : neutrophils ≥1.5× L09 /L, platelets ≥100×109/L, hemoglobin ≥90g/L; II. Liver function: ALT and AST, ALT and AST≤3×ULN in patients without liver metastasis, ALT and AST≤5×ULN in patients with liver metastasis;Total bilirubin (TBil) ≤1.5×ULN (Gilbert syndrome patients, ≤3 ×ULN); Iii. Renal function: Serum creatinine (CR) ≤1.5×ULN or creatinine clearance (CCR) ≥50ml/ min (subjects receiving carboplatin) or ≥60ml/ min (subjects receiving cisplatin); IV. Coagulation function: APTT, INR, PT ≤1.5×ULN; V. Echocardiography: left ventricular ejection fraction (LVEF) ≥50%; 10) Women should agree to use contraceptives (such as intrauterine devices [IUDs], contraceptives or condoms) during the study period and for 6 months after the end of the study;Negative blood pregnancy test within 7 days prior to study enrolment and must be non-lactating;Men should agree to use contraception during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

* 1) The patient had necrotic lesions and was judged by the investigator to be at risk of massive bleeding; 2) A history of hypersensitivity to amlotinib or pabrizumab or any excipients; 3) Previous use of antiangiogenic drugs (such as amlotinib, apatinib, bevacizumab, Endox, etc.); 4) The patient is using (or cannot be discontinued within 1 week prior to the first dosing of the study treatment) a Chinese herbal medicine indicated for antitumor use; 5) poorly controlled pleural effusion, pericardial effusion or ascites requiring frequent drainage;Patients with indwelling catheters (such as the Pleurx ® catheter) are allowed to participate; 6) At the beginning of study treatment, there was still an uncured toxic reaction from previous treatment and CTCAE 5.0 was higher than level 1 (except for alopecia); 7) Spinal cord compression or symptomatic untreated brain or spinal cord metastases (except asymptomatic, stable condition, and no need for steroid therapy for 4 weeks prior to study treatment); 8) poorly controlled tumor-related pain.Patients who require analgesics must receive a steady dose before entering the study.Symptomatic lesions suitable for palliative radiotherapy (e.g., bone metastases or metastases leading to nerve damage) should be treated before enrolment.Prior to enrolment, local-regional treatment of asymptomatic metastatic lesions with further growth that may result in functional deficits or intractable pain (e.g., epidural metastases currently not associated with spinal cord compression) should be considered, if appropriate.

  9) Hepatitis B, hepatitis C or human immunodeficiency virus (HIV antibody positive).Patients with positive hepatitis B antibodies were only eligible to participate in the study if they had HBV DNA ˂2000cps/ml.Patients with hepatitis C antibody positive were eligible to participate in the study only if polymerase chain reaction showed HCV RNA negative; 10) Randomization of malignancies other than advanced head and neck squamous cell carcinoma with negligible risk of metastasis or death and expected radical outcome after treatment within the first 5 years (e.g.,Adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer for radical treatment, and ductal carcinoma in situ for radical surgery); 11) Had major surgery other than a diagnosis of advanced head and neck squamous cell carcinoma within 28 days prior to randomization or was expected to require major surgery during the study period; 12) patients who have had previous bone marrow transplantation or previous solid organ transplantation; 13) Any live vaccine (for example, vaccines against infectious diseases, such as influenza, varicella, etc.) was given within the first 4 weeks (28 days) of randomization; 14) any factors that may affect the patient's oral administration, such as inability to swallow, post-gastrointestinal resection, chronic diarrhea, and intestinal obstruction; 15) Meets any of the following cardiac criteria: mean corrected QT interval (QTc) from an electrocardiogram (ECG) in the resting state;470 msec (for the first anomaly, the test was retest once within 48 h, calculated based on the average result of two times).A variety of clinically significant cardiac rhythm, conduction, and resting ECG abnormalities, such as complete left bundle branch block, degree III, degree II, PR interval >250 msec.Various factors that may increase the risk of prolonged QTC or arrhythmic events, such as coronary heart disease, heart failure, hypokalemia, congenital long QT syndrome, a family history of first-degree relative with long QT syndrome or sudden unexplained death under age 40, and being on any known medication for prolonged QT; 16) Patients with any severe and/or uncontrolled disease, including but not limited to: patients with poor blood pressure control (systolic > 150 mmHg, diastolic > 100 mmHg);Suffer from myocardial ischemia or myocardial infarction, arrhythmias (including QTc ≥440ms) and congestive heart failure (New York Heart Association (NYHA) grade) of grade I or above;Active or uncontrolled severe infection (≥CTC AE grade 2 infection);Cirrhosis, decompensated liver disease;Renal failure requires hemodialysis or peritoneal dialysis;Poor diabetes control (fasting blood glucose (FBG) > 10mmol/L);Routine urine indicated urinary protein ≥++, and confirmed 24-hour urinary protein quantitative > 1.0 g; 17) Patients with epileptic seizures requiring treatment, with a history of psychotropic substance abuse and unable to quit or with mental disorders; 18) Previous history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonia requiring steroid treatment, and clinically evidenced active interstitial lung disease; 19) thrombotic or embolic venous or arterial events, such as cerebrovascular accidents, including transient ischemic attack, arterial thrombosis, deep vein thrombosis and pulmonary embolism, occurred within 6 months before enrollment;Has a history of hemorrhagic disease or abnormal blood clotting.

  20) Lactating female patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-18 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
objective response rates(ORR) | 1 year
  To evaluate objective response rates of first-line Pembrolizumab combined with Anlotinib in Chinese patients with recurrent and/or metastatic head and neck squamous cell carcinoma (HNSCC) with PD-L1 CPS≥1

SECONDARY OUTCOMES:
disease control rate(DCR) | 3 year
  To evaluate other efficacy indicators of first-line Pembrolizumab combined with Anlotinib in Chinese patients with recurrent and/or metastatic head and neck squamous cell carcinoma with PD-L1 CPS≥1, including disease control rate(DCR)
duration of response(DOR) | 3 year
  To evaluate other efficacy indicators of first-line Pembrolizumab combined with Anlotinib in Chinese patients with recurrent and/or metastatic head and neck squamous cell carcinoma with PD-L1 CPS≥1, duration of response(DOR)
progression-free survival(PFS) | 3 year
  To evaluate other efficacy indicators of first-line Pembrolizumab combined with Anlotinib in Chinese patients with recurrent and/or metastatic head and neck squamous cell carcinoma with PD-L1 CPS≥1, progression-free survival(PFS)
overall survival (OS) | 5 year
  To evaluate other efficacy indicators of first-line Pembrolizumab combined with Anlotinib in Chinese patients with recurrent and/or metastatic head and neck squamous cell carcinoma with PD-L1 CPS≥1, overall survival (OS)

OTHER OUTCOMES:
tumor mutation burden（TMB） | 3 year
  Correlation results of tumor mutation burden（TMB）
T cell gene expression | 3 year
  Correlation results of T cell gene expression

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, Principal Investigator — Cancer Institute/Hospital, Chinese Academy of Medical Sciences&Peking Union Medical college
Locations (1):
- National Cancer Center/Cancer Hospitial,Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No